CLINICAL TRIAL: NCT04056676
Title: Analgesic Effect of Adding Thoracic Paravertebral Nerve Blocks to Modified PEC Block in Breast Cancer Surgery, Prospective Randomized Controlled Study
Brief Title: Analgesic Effect of Adding Thoracic Paravertebral Nerve Blocks to Modified PEC Block in Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Assistant professor, Department of Anesthesiology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SI 475/2019
Record Dates: First submitted 2019-08-08; First posted 2019-08-14 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer Female; Pain, Postoperative
Keywords: Postoperative pain; Thoracic paravertebral block; Modified PEC block; Breast cancer; Total mastectomy with sentinel lymph node clearance
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: group A Intraoperative modified PEC block only group B Preoperative thoracic paravertebral block plus intraoperative modified PEC block
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomized group of patient is identified and sealed in envelope. There is not written group in anesthetic record. Postoperative outcomes are assessed by Acute Pain Service nurse or a resident (co-investigator who blinds to the technique).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraoperative modified PEC block only (Active Comparator): Intraoperative modified PEC block with 0.5% bupivacaine 20 ml plus adrenaline 100 ug by surgeon
  Interventions: Procedure: Intraoperative modified PEC block; Procedure: GA with ETT
- Adding preoperative thoracic paravertebral nerve block (Experimental): Preoperative thoracic paravertebral nerve block with 0.5% bupivacaine 20 ml plus adrenaline 100 ug and intraoperative modified PEC block with 0.5% bupivacaine 20 ml plus adrenaline 100 ug by surgeon
  Interventions: Procedure: Thoracic paravertebral block under ultrasound guidance; Procedure: Intraoperative modified PEC block; Procedure: GA with ETT

INTERVENTIONS:
Procedure: Thoracic paravertebral block under ultrasound guidance — Ultrasound-guided thoracic paravertebral blocks in T2, T4 level
  Other Names: USG-TPVB
  Arms: Adding preoperative thoracic paravertebral nerve block
Procedure: Intraoperative modified PEC block — Pectoral nerve block by surgeon under direct vision after total mastectomy
  Other Names: Modified PEC block
Procedure: GA with ETT — General anesthesia with endotracheal intubation

SUMMARY:
To compare efficacy and safety of adding thoracic paravertebral nerve blocks to modified PEC block versus modified PEC block only in breast cancer surgery. This study evaluate systemic opioid requirement in 48 hours in primary outcome and the analgesic profile ( pain score at rest and on shoulder movement), opioid-related side effects and nerve blocks complications.

DETAILED DESCRIPTION:
Regional anesthesia has been used and studied extensively in breast surgery as an opioid-sparing strategy, with block of the intercostal supply by thoracic paravertebral block (TPVB) becoming a popular technique.

This prospective randomized controlled trial is aimed to study the proper regional nerve block technique to reach the postoperative opioid-free requirement modality for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) grade I-III
* Aged ≥ 18-80 years old
* Elective unilateral total mastectomy with sentinel lymph node biopsy or lymph node dissection

Exclusion Criteria:

* Patient refusal
* Language barrier or inability to communicate with the operating team
* Allergy to local anesthetic
* Bleeding disorder
* Previous breast surgery or thoracic radiation therapy
* BMI ≥ 30
* Patient who can not understand the proper use of intravenous patient-controlled analgesia machine or who has the problem with communication
* Chronic pain patient

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative fentanyl consumption | at postoperative 24 hours
  Cumulative fentanyl consumption within postoperative 24 hours
Postoperative fentanyl consumption | at postoperative 48 hours
  Cumulative fentanyl consumption within postoperative 24-48 hours

SECONDARY OUTCOMES:
Intraoperative fentanyl use | Intraoperation
  Dosage of intraoperative fentanyl usage in micrograms
Postoperative pain score at rest | at postoperative 0 hour (PACU arrival)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | at postoperative 30 min (in PACU)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | at postoperative 1 hour (in PACU)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | Postoperative 6 hour (at ward)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | Postoperative 12 hour (at ward)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | Postoperative 18 hour (at ward)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score at rest | Postoperative 24 hour (at ward)
  Numeric rating score 0-10 (0= no pain, 10= worst pain imaginable)
Postoperative pain score on shoulder movement | Postoperative 1 hour (at PACU)
  Numeric rating score ((0= no pain, 10= worst pain imaginable)
Postoperative pain score on shoulder movement | Postoperative first day (at ward)
  Numeric rating score ((0= no pain, 10= worst pain imaginable)
Postoperative pain score on shoulder movement | Postoperative second day (at ward)
  Numeric rating score ((0= no pain, 10= worst pain imaginable)
First time to fentanyl requirement by IV PCA | Within 24 hours
  time to require fentanyl patient-controlled intravenous analgesia
Percentage of patients presenting with opioid-related adverse effects | Within 48 hours
  adverse effects include postoperative nausea, vomiting, dizziness, pruritus
Percentage of patients presenting with nerve block complications | Within 48 hours
  nerve block complications include pneumothorax, hypotension, local anesthetic systemic toxicity, Horner syndrome
Length of hospital stay | From preoperative admission until hospital discharge
  Number of hospital admission days
Patient's satisfaction scale score | At postoperative 48 hours
  Satisfaction scale score 0-10 (0= highly unsatisfied, 10= highly satisfied)
Cost effectiveness analysis | Within 48 hours
  Cost of adding nerve block and postoperative pain score

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Background] Missair A, Cata JP, Votta-Velis G, Johnson M, Borgeat A, Tiouririne M, Gottumukkala V, Buggy D, Vallejo R, Marrero EB, Sessler D, Huntoon MA, Andres J, Casasola OL. Impact of perioperative pain management on cancer recurrence: an ASRA/ESRA special article. Reg Anesth Pain Med. 2019 Jan;44(1):13-28. doi: 10.1136/rapm-2018-000001. PMID 30640648
- [Background] Woodworth GE, Ivie RMJ, Nelson SM, Walker CM, Maniker RB. Perioperative Breast Analgesia: A Qualitative Review of Anatomy and Regional Techniques. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):609-631. doi: 10.1097/AAP.0000000000000641. PMID 28820803
- [Background] Wynne R, Lui N, Tytler K, Koffsovitz C, Kirwa V, Riedel B, Ryan S. The Trajectory of Postoperative Pain Following Mastectomy with and without Paravertebral Block. Pain Manag Nurs. 2017 Aug;18(4):234-242. doi: 10.1016/j.pmn.2017.03.003. Epub 2017 Jun 7. PMID 28601480
- [Background] Syal K, Chandel A. Comparison of the post-operative analgesic effect of paravertebral block, pectoral nerve block and local infiltration in patients undergoing modified radical mastectomy: A randomised double-blind trial. Indian J Anaesth. 2017 Aug;61(8):643-648. doi: 10.4103/ija.IJA_81_17. PMID 28890559
- [Background] Terkawi AS, Tsang S, Sessler DI, Terkawi RS, Nunemaker MS, Durieux ME, Shilling A. Improving Analgesic Efficacy and Safety of Thoracic Paravertebral Block for Breast Surgery: A Mixed-Effects Meta-Analysis. Pain Physician. 2015 Sep-Oct;18(5):E757-80. PMID 26431130
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971